CLINICAL TRIAL: NCT00006890
Title: A Randomized Phase II Dose Finding Study Of Thalidomide And Prednisone As Maintenance Therapy Following Autologous Stem Cell Transplant In Patients With Multiple Myeloma
Brief Title: Thalidomide and Prednisone Following Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MY9; CAN-NCIC-MY9 (Other: PDQ); CELGENE-CAN-NCIC-MY9 (Other: Celgene); CDR0000068337 (Other: PDQ)
Record Dates: First submitted 2000-12-06; First posted 2004-03-08 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Prednisone; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prednisone plus Thalidomide (Experimental): After Autologous Stem Cell Infusion
  Interventions: Drug: prednisone; Drug: thalidomide

INTERVENTIONS:
Drug: prednisone — Prednisone 50mg on alternate days
Drug: thalidomide — THALIDOMIDE 200 mg qhs

SUMMARY:
RATIONALE: Thalidomide may stop the growth of multiple myeloma by stopping blood flow to the tumor. Prednisone may be effective in preventing relapse of multiple myeloma.

PURPOSE: Randomized phase II trial to compare the effectiveness of two doses of thalidomide combined with prednisone following peripheral stem cell transplantation in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine which dose of thalidomide (200 mg vs 400 mg) combined with prednisone is the optimally tolerated dose when used as maintenance therapy following autologous stem cell transplantation in patients with multiple myeloma. II. Compare the response rate in patients treated with these regimens. III. Compare the progression-free and overall survival in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to age (60 and over vs under 60). Within 60-100 days after autologous stem cell transplantation, patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive lower dose oral thalidomide daily and oral prednisone every other day. Arm II: Patients receive higher dose thalidomide daily and oral prednisone every other day. Treatment continues for 2 years in the absence of disease progression or unacceptable toxicity. Patients are followed monthly for 6 months, every 3 months, and then at time of disease progression.

PROJECTED ACCRUAL: A total of 40-80 patients (20-40 per arm) will be accrued for this study within 17-21 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven multiple myeloma Initial diagnosis must have been confirmed by one of the following prior to initial treatment for multiple myeloma: Biopsy of an osteolytic lesion or soft tissue tumor composed of plasma cells Bone marrow aspirate and/or biopsy demonstrating at least 10% plasmacytosis Bone marrow containing less than 10% plasma cells but with at least 1 bony lesion and the M-protein criteria outlined below Measurable serum M-component of IgG, IgA, IgD, or IgE at initial diagnosis OR If only light chain disease (urine M-protein only) present, then the urinary excretion of light chain (Bence Jones) protein must have been at least 1.0 g/24 hours at time of initial diagnosis Must have undergone autologous stem cell transplantation within 1 year of beginning initial chemotherapy for multiple myeloma Must be randomized 60-100 days after autologous stem cell infusion No evidence of progressive disease

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-2 Life expectancy: At least 6 months Hematopoietic: See Disease Characteristics Granulocyte count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: AST and/or ALT no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 1.5 times ULN Renal: Creatinine no greater than 3 times ULN Cardiovascular: No uncontrolled hypertension Other: Not pregnant or nursing Negative pregnancy test Fertile female patients must use 2 effective methods of contraception (1 barrier and 1 hormonal) during and for 1 month after study Fertile male patients must use effective barrier contraception during and for 1 month after study No other medical condition that would preclude long term use of prednisone or thalidomide No other malignancy within the past 5 years except adequately treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix No diabetes with end stage organ damage No history of gastric ulceration or bleeding No avascular necrosis of the hips No peripheral neuropathy causing symptomatic dysfunction Sensory symptoms induced by vincristine allowed No demonstrated hypersensitivity to thalidomide or its components No other major medical illness that would increase risk or preclude study No employment that prohibits the use of sedatives (due to known effect of thalidomide)

PRIOR CONCURRENT THERAPY: Biologic: See Disease Characteristics No prior thalidomide Chemotherapy: See Disease Characteristics Endocrine: Not specified Radiotherapy: Not specified Surgery: Not specified Other: No other concurrent anticancer treatment No other concurrent investigational therapy

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2000-07-12 (Actual); Primary Completion 2002-05-03 (Actual); Study Completion 2008-12-15 (Actual)

PRIMARY OUTCOMES:
incidence of drop-out or dose reduction | 2 years
  incidence of drop-out or dose reduction due to toxicity within 6 months from the start of treatment.

SECONDARY OUTCOMES:
Response rate | 2 years
Time to progression | 2 years
Overall survival | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: A. Keith Stewart, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (64):
- St. Mary's/Duluth Clinic Health System, Duluth, Minnesota, United States
- Canada (63):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Lethbridge Cancer Clinic, Lethbridge, Alberta
  - Burnaby Hospital Regional Cancer Centre, Burnaby, British Columbia
  - Nanaimo Cancer Clinic, Nanaimo, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - St. Paul's Hospital - Vancouver, Vancouver, British Columbia
  - G. Steinhoff Clinical Research, Victoria, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cape Breton Cancer Centre, Sydney, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Hamilton and Disrict Urology Association, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - York County Hospital, Newmarket, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Male Health Centre/CMX Research Inc., Oakville, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Scarborough Hospital - General Site, Scarborough Village, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Women's College Campus, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier Regional de Lanaudiere, Joliette, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier de l'Universite' de Montreal, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Kells Medical Research Group Inc., Pointe-Claire, Quebec
  - CHU de Quebec - L'Hotel-Dieu de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - Centre Hospitalier Regional de Rimouski, Rimouski, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Lions Gate Hospital, North Vancouver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stewart AK, Chen CI, Howson-Jan K, White D, Roy J, Kovacs MJ, Shustik C, Sadura A, Shepherd L, Ding K, Meyer RM, Belch AR. Results of a multicenter randomized phase II trial of thalidomide and prednisone maintenance therapy for multiple myeloma after autologous stem cell transplant. Clin Cancer Res. 2004 Dec 15;10(24):8170-6. doi: 10.1158/1078-0432.CCR-04-1106. PMID 15623591
- [Result] Stewart KA, Chen C, Howson-Jan K, et al.: A randomized phase II dose-finding trial of thalidomide and prednisone as maintenance therapy for myeloma following autologous stem cell transplant. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1073, 2002.